CLINICAL TRIAL: NCT06116110
Title: A Prospective, Observational, Long-term Follow-up Study for Subjects Who Previously Received Zamtocabtagene Autoleucel in a United States Miltenyi Biomedicine-Sponsored Clinical Study
Brief Title: Lentiviral Gene Therapy (Zamtocabtagene Autoleucel) LTFU
Status: Recruiting | Type: Observational
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: M-2023-401
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Chimeric antigen receptor; CAR T; CD19; CD20
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-term Follow-Up: No intervention
  Interventions: Other: Long-term Follow-Up

INTERVENTIONS:
Other: Long-term Follow-Up — No intervention

SUMMARY:
This is an observational long-term follow-up (LTFU) study for subjects who previously received zamtocabtagene autoleucel, known as MB-CART2019.1.

DETAILED DESCRIPTION:
This is a non-therapeutic study design. After successful screening, subjects will be monitored for potential gene therapy-related adverse events for up to 15 years post MB-CART2019.1 infusion. Subjects will be assessed yearly for the occurrence of delayed adverse events (AEs), monitored for replication competent lentivirus (RCL) and assessed for long term efficacy as well as CAR-T persistence.

ELIGIBILITY:
Inclusion Criteria:

* Received zamtocabtagene autoleucel in a Miltenyi Biomedicine-sponsored clinical study and have either completed the study or have discontinued early from the study.
* Provided written informed consent to participate in this study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received MB-CART2019.1
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2039-12-01 (Estimated); Study Completion 2039-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of serious and non serious adverse events of special interest | Up to 15 years
  AESIs will be collected

SECONDARY OUTCOMES:
Number of subjects with measurable replication competent lentivirus in peripheral blood (if positive at study entry) | Up to 15 years
  Peripheral blood samples may be collected for RCL assessment
Duration of zamtocabtagene autoleucel persistence | Up to 5 years
  Peripheral blood samples will be collected to test for CAR T cells
Objective response rate | Up to 15 years
  ORR
Overall Survival | Up to 15 years
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Remi Kaleta, MD, Study Director — Miltenyi Biomedicine GmbH
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - University of Maryland Marlene and Stewart Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin